CLINICAL TRIAL: NCT03783091
Title: A Phase II Double Blind Randomized Controlled Trial of High Dose Vitamin B12 in Septic Shock
Brief Title: A Trial of Vitamin B12 in Septic Shock
Acronym: B12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jayshil J. Patel, MD, Associate Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32950
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Hydroxocobalamin; Vitamin B 12; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Vitamin B12a is bright red and excreted in the urine. Due to this, patient allocation cannot be masked for patients or individuals who may care for them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydroxocobalamin (Experimental): Single IV infusion administered over a 10-15 minute period
  Interventions: Drug: Hydroxocobalamin
- Saline Placebo (Placebo Comparator): Single IV saline administered over a 10-15 minute period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxocobalamin — Single IV administration of Vitamin B12
  Other Names: Cyanokit
  Arms: Hydroxocobalamin
Drug: Placebo — Single IV administration of saline
  Other Names: 200-250 mL of intravenous saline or dextrose
  Arms: Saline Placebo

SUMMARY:
This study will randomize 20 septic shock patients to receive either a single 5 gram dose of IV vitamin B12 (Cyanokit® Meridian Medical Technologies, Columbia, MD) versus placebo in addition to standard of care to test the feasibility of completing clinical and laboratory protocols.

DETAILED DESCRIPTION:
Following informed consent from patient's legally authorized representative, patients will be randomized to hydroxocobalamin or saline. Patients will have blood samples drawn up to 3 hours pre-dose and 3 hours post-dose to measure for hydrogen sulfide levels. Patients will also be followed for 3 hours after study drug infusion to monitor and record vasopressor dependence in norepinephrine-equivalent dose. Patients will then be followed through their medical record for 28 days to determine persistent organ dysfunction syndrome (PODS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at least 18 years of age
* Admitted to the Medical Intensive Care Unit (MICU) service at Froedtert Hospital
* Diagnosis of septic shock, as defined by sepsis-3 criteria

Exclusion Criteria:

* History of calcium oxaluria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of completing clinical and laboratory protocols | 28 days
  Feasibility of completing clinical and laboratory protocols

SECONDARY OUTCOMES:
Hydrogen Sulfide Concentration | 3 hours
  Difference between pre- and post-dose hydrogen sulfide levels
Persistent Organ Dysfunction Syndrome (PODS) | 28 days
  Prevalence of Persistent organ dysfunction syndrome (PODS)
Change in vasopressor dose | 3, 24, and 48 hours
  Vasopressor dose in mcg/kg/min (norepinephrine equivelents)
Mortality | 28 days
  Intensive care unit and hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jayshil J Patel, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Abraham E, Reinhart K, Svoboda P, Seibert A, Olthoff D, Dal Nogare A, Postier R, Hempelmann G, Butler T, Martin E, Zwingelstein C, Percell S, Shu V, Leighton A, Creasey AA. Assessment of the safety of recombinant tissue factor pathway inhibitor in patients with severe sepsis: a multicenter, randomized, placebo-controlled, single-blind, dose escalation study. Crit Care Med. 2001 Nov;29(11):2081-9. doi: 10.1097/00003246-200111000-00007. PMID 11700399
- [Background] Bernard GR, Wheeler AP, Russell JA, Schein R, Summer WR, Steinberg KP, Fulkerson WJ, Wright PE, Christman BW, Dupont WD, Higgins SB, Swindell BB. The effects of ibuprofen on the physiology and survival of patients with sepsis. The Ibuprofen in Sepsis Study Group. N Engl J Med. 1997 Mar 27;336(13):912-8. doi: 10.1056/NEJM199703273361303. PMID 9070471
- [Background] Lopez A, Lorente JA, Steingrub J, Bakker J, McLuckie A, Willatts S, Brockway M, Anzueto A, Holzapfel L, Breen D, Silverman MS, Takala J, Donaldson J, Arneson C, Grove G, Grossman S, Grover R. Multiple-center, randomized, placebo-controlled, double-blind study of the nitric oxide synthase inhibitor 546C88: effect on survival in patients with septic shock. Crit Care Med. 2004 Jan;32(1):21-30. doi: 10.1097/01.CCM.0000105581.01815.C6. PMID 14707556
- [Background] Lorente JA, Landin L, De Pablo R, Renes E, Liste D. L-arginine pathway in the sepsis syndrome. Crit Care Med. 1993 Sep;21(9):1287-95. doi: 10.1097/00003246-199309000-00010. PMID 8370291
- [Background] Szakmany T, Hauser B, Radermacher P. N-acetylcysteine for sepsis and systemic inflammatory response in adults. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD006616. doi: 10.1002/14651858.CD006616.pub2. PMID 22972094
- [Background] Takala J, Ruokonen E, Webster NR, Nielsen MS, Zandstra DF, Vundelinckx G, Hinds CJ. Increased mortality associated with growth hormone treatment in critically ill adults. N Engl J Med. 1999 Sep 9;341(11):785-92. doi: 10.1056/NEJM199909093411102. PMID 10477776
- [Background] Shatalin K, Shatalina E, Mironov A, Nudler E. H2S: a universal defense against antibiotics in bacteria. Science. 2011 Nov 18;334(6058):986-90. doi: 10.1126/science.1209855. PMID 22096201
- [Background] Lambden S, Creagh-Brown BC, Hunt J, Summers C, Forni LG. Definitions and pathophysiology of vasoplegic shock. Crit Care. 2018 Jul 6;22(1):174. doi: 10.1186/s13054-018-2102-1. PMID 29980217
- [Background] Kosir M, Podbregar M. Advances in the Diagnosis of Sepsis: Hydrogen Sulfide as a Prognostic Marker of Septic Shock Severity. EJIFCC. 2017 May 1;28(2):134-141. eCollection 2017 May. PMID 28757821
- [Background] Zhang H, Moochhala SM, Bhatia M. Endogenous hydrogen sulfide regulates inflammatory response by activating the ERK pathway in polymicrobial sepsis. J Immunol. 2008 Sep 15;181(6):4320-31. doi: 10.4049/jimmunol.181.6.4320. PMID 18768890
- [Background] Goslar T, Mars T, Podbregar M. Total plasma sulfide as a marker of shock severity in nonsurgical adult patients. Shock. 2011 Oct;36(4):350-5. doi: 10.1097/SHK.0b013e31822bcfd0. PMID 21897337
- [Background] Li L, Bhatia M, Zhu YZ, Zhu YC, Ramnath RD, Wang ZJ, Anuar FB, Whiteman M, Salto-Tellez M, Moore PK. Hydrogen sulfide is a novel mediator of lipopolysaccharide-induced inflammation in the mouse. FASEB J. 2005 Jul;19(9):1196-8. doi: 10.1096/fj.04-3583fje. Epub 2005 Apr 29. PMID 15863703
- [Background] Zundel MT, Feih JT, Rinka JRG, Boettcher BT, Freed JK, Kaiser M, Ghadiali HY, Tawil JN, Woehlck HJ, Pagel PS. Hydroxocobalamin With or Without Methylene Blue May Improve Fluid Balance in Critically Ill Patients With Vasoplegic Syndrome After Cardiac Surgery: A Report of Two Cases. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):452-457. doi: 10.1053/j.jvca.2017.04.002. Epub 2017 Apr 5. No abstract available. PMID 28778773
- [Background] Truong DH, Mihajlovic A, Gunness P, Hindmarsh W, O'Brien PJ. Prevention of hydrogen sulfide (H2S)-induced mouse lethality and cytotoxicity by hydroxocobalamin (vitamin B(12a)). Toxicology. 2007 Dec 5;242(1-3):16-22. doi: 10.1016/j.tox.2007.09.009. Epub 2007 Sep 15. PMID 17976885
- [Background] Brenner M, Benavides S, Mahon SB, Lee J, Yoon D, Mukai D, Viseroi M, Chan A, Jiang J, Narula N, Azer SM, Alexander C, Boss GR. The vitamin B12 analog cobinamide is an effective hydrogen sulfide antidote in a lethal rabbit model. Clin Toxicol (Phila). 2014 Jun;52(5):490-7. doi: 10.3109/15563650.2014.904045. Epub 2014 Apr 9. PMID 24716792
- [Background] Ng PC, Hendry-Hofer TB, Garrett N, Brenner M, Mahon SB, Maddry JK, Haouzi P, Boss GR, Gibbons TF, Arana AA, Bebarta VS. Intramuscular cobinamide versus saline for treatment of severe hydrogen sulfide toxicity in swine. Clin Toxicol (Phila). 2019 Mar;57(3):189-196. doi: 10.1080/15563650.2018.1504955. Epub 2018 Nov 15. PMID 30430872
- [Background] Weinberg JB, Chen Y, Jiang N, Beasley BE, Salerno JC, Ghosh DK. Inhibition of nitric oxide synthase by cobalamins and cobinamides. Free Radic Biol Med. 2009 Jun 15;46(12):1626-32. doi: 10.1016/j.freeradbiomed.2009.03.017. Epub 2009 Mar 27. PMID 19328848
- [Background] Zhang H, Zhi L, Moochhala S, Moore PK, Bhatia M. Hydrogen sulfide acts as an inflammatory mediator in cecal ligation and puncture-induced sepsis in mice by upregulating the production of cytokines and chemokines via NF-kappaB. Am J Physiol Lung Cell Mol Physiol. 2007 Apr;292(4):L960-71. doi: 10.1152/ajplung.00388.2006. Epub 2007 Jan 5. PMID 17209138
- [Background] An SS, Henson CP, Freundlich RE, McEvoy MD. Case report of high-dose hydroxocobalamin in the treatment of vasoplegic syndrome during liver transplantation. Am J Transplant. 2018 Jun;18(6):1552-1555. doi: 10.1111/ajt.14736. Epub 2018 Apr 2. PMID 29573551
- [Background] Woehlck HJ, Boettcher BT, Lauer KK, Cronin DC, Hong JC, Zimmerman MA, Kim J, Selim M. Hydroxocobalamin for Vasoplegic Syndrome in Liver Transplantation: Restoration of Blood Pressure Without Vasospasm. A A Case Rep. 2016 Dec 15;7(12):247-250. doi: 10.1213/XAA.0000000000000398. PMID 27749291
- [Background] Boettcher BT, Woehlck HJ, Reck SE, Hong JC, Zimmerman MA, Kim J, Zundel MT, Freed JK, Pagel PS. Treatment of Vasoplegic Syndrome With Intravenous Hydroxocobalamin During Liver Transplantation. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1381-1384. doi: 10.1053/j.jvca.2016.10.011. Epub 2016 Oct 14. No abstract available. PMID 28012726
- [Background] Burnes ML, Boettcher BT, Woehlck HJ, Zundel MT, Iqbal Z, Pagel PS. Hydroxocobalamin as a Rescue Treatment for Refractory Vasoplegic Syndrome After Prolonged Cardiopulmonary Bypass. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):1012-1014. doi: 10.1053/j.jvca.2016.08.019. Epub 2016 Aug 18. No abstract available. PMID 27838199
- [Background] Shah PR, Reynolds PS, Pal N, Tang D, McCarthy H, Spiess BD. Hydroxocobalamin for the treatment of cardiac surgery-associated vasoplegia: a case series. Can J Anaesth. 2018 May;65(5):560-568. doi: 10.1007/s12630-017-1029-3. Epub 2017 Dec 5. PMID 29209927
- [Background] Modis K, Bos EM, Calzia E, van Goor H, Coletta C, Papapetropoulos A, Hellmich MR, Radermacher P, Bouillaud F, Szabo C. Regulation of mitochondrial bioenergetic function by hydrogen sulfide. Part II. Pathophysiological and therapeutic aspects. Br J Pharmacol. 2014 Apr;171(8):2123-46. doi: 10.1111/bph.12368. PMID 23991749
- [Background] Bice JS, Jones BR, Chamberlain GR, Baxter GF. Nitric oxide treatments as adjuncts to reperfusion in acute myocardial infarction: a systematic review of experimental and clinical studies. Basic Res Cardiol. 2016 Mar;111(2):23. doi: 10.1007/s00395-016-0540-y. Epub 2016 Feb 24. PMID 26912064
- [Background] Ozaki KS, Kimura S, Murase N. Use of carbon monoxide in minimizing ischemia/reperfusion injury in transplantation. Transplant Rev (Orlando). 2012 Apr;26(2):125-39. doi: 10.1016/j.trre.2011.01.004. Epub 2011 Oct 13. PMID 22000659
- [Background] Eckstein M. Enhancing public health preparedness for a terrorist attack involving cyanide. J Emerg Med. 2008 Jul;35(1):59-65. doi: 10.1016/j.jemermed.2007.03.040. Epub 2007 Aug 29. PMID 17976798
- [Background] Anseeuw K, Delvau N, Burillo-Putze G, De Iaco F, Geldner G, Holmstrom P, Lambert Y, Sabbe M. Cyanide poisoning by fire smoke inhalation: a European expert consensus. Eur J Emerg Med. 2013 Feb;20(1):2-9. doi: 10.1097/MEJ.0b013e328357170b. PMID 22828651
- [Background] Khanna A, English SW, Wang XS, Ham K, Tumlin J, Szerlip H, Busse LW, Altaweel L, Albertson TE, Mackey C, McCurdy MT, Boldt DW, Chock S, Young PJ, Krell K, Wunderink RG, Ostermann M, Murugan R, Gong MN, Panwar R, Hastbacka J, Favory R, Venkatesh B, Thompson BT, Bellomo R, Jensen J, Kroll S, Chawla LS, Tidmarsh GF, Deane AM; ATHOS-3 Investigators. Angiotensin II for the Treatment of Vasodilatory Shock. N Engl J Med. 2017 Aug 3;377(5):419-430. doi: 10.1056/NEJMoa1704154. Epub 2017 May 21. PMID 28528561
- [Background] Shen X, Peter EA, Bir S, Wang R, Kevil CG. Analytical measurement of discrete hydrogen sulfide pools in biological specimens. Free Radic Biol Med. 2012 Jun 1-15;52(11-12):2276-83. doi: 10.1016/j.freeradbiomed.2012.04.007. Epub 2012 Apr 19. PMID 22561703
- [Background] Puskarich MA, Kline JA, Watts JA, Shirey K, Hosler J, Jones AE. Early alterations in platelet mitochondrial function are associated with survival and organ failure in patients with septic shock. J Crit Care. 2016 Feb;31(1):63-7. doi: 10.1016/j.jcrc.2015.10.005. Epub 2015 Oct 26. PMID 26511963
- [Derived] Patel JJ, Willoughby R, Peterson J, Carver T, Zelten J, Markiewicz A, Spiegelhoff K, Hipp LA, Canales B, Szabo A, Heyland DK, Stoppe C, Zielonka J, Freed JK. High-Dose IV Hydroxocobalamin (Vitamin B12) in Septic Shock: A Double-Blind, Allocation-Concealed, Placebo-Controlled Single-Center Pilot Randomized Controlled Trial (The Intravenous Hydroxocobalamin in Septic Shock Trial). Chest. 2023 Feb;163(2):303-312. doi: 10.1016/j.chest.2022.09.021. Epub 2022 Sep 26. PMID 36174744